CLINICAL TRIAL: NCT03824483
Title: Phase 2 Study of Zanubrutinib, Obinutuzumab, and Venetoclax in Previously Untreated Patients With Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL) and Mantle Cell Lymphoma (MCL)
Brief Title: Study of Zanubrutinib, Obinutuzumab, and Venetoclax in Patients With Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Leukemia (SLL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: BeiGene USA, Inc. (Industry); Roche-Genentech (Industry); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-427
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Leukemia (SLL)
Keywords: Zanubrutinib; Obinutuzumab; Venetoclax; 18-427
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib; obinutuzumab; venetoclax

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled in a single-stage phase 2 design.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BOVEN regimen (Experimental): Patients will be given zanubrutinib (160mg by mouth BID) and obinutuzumab (1000mg IVPB on Days 1*, 8 and 15 of Cycle 1 and on Day 1 of Cycles 2 through 8) starting on Cycle 1 (28-day cycles). * On Cycle 1, obinituzumab will be administered in "split dose" at 100mg IVPB on Day 1 and 900mg IVPB on Day 2 in patients at increased risk for IRR (ALC >25,000 cells/ul or baseline lymph nodes >5 cm diameter). Venetoclax will be added to the regimen starting on Cycle 3, and will be incorporated into the regimen using the 5-week ramp-up schedule to mitigate the risk of tumor lysis syndrome (beginning at 20mg and gradually increasing to 400mg), and venetoclax will be administered a ta fixed dose level of 400mg by mouth daily of 28-day cycles thereafter.
  Interventions: Drug: Zanubrutinib; Drug: Obinutuzumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Zanubrutinib — zanubrutinib (160mg by mouth BID)
Drug: Obinutuzumab — obinutuzumab (1000mg IVPB on Days 1*, 8 and 15 of Cycle 1 and on Day 1 of Cycles 2 through 8) starting on Cycle 1 (28-day cycles). * On Cycle 1, obinituzumab will be administered in "split dose" at 100mg IVPB on Day 1 and 900mg IVPB on Day 2 in patients at increased risk for IRR (ALC >25,000 cells/ul or baseline lymph nodes >5 cm diameter).
  Other Names: GA101
Drug: Venetoclax — Venetoclax will be added to the regimen starting on Cycle 3, and will be incorporated into the regimen using the 5-week ramp-up schedule to mitigate the risk of tumor lysis syndrome (beginning at 20mg and gradually increasing to 400mg), and venetoclax will be administered a ta fixed dose level of 400mg by mouth daily of 28-day cycles thereafter.
  Other Names: ABT-199

SUMMARY:
The purpose of this study is to determine the rate of minimum residual disease (MRD) negative response (i.e. the rate of no evidence of disease) of the study drugs, zanubrutinib, obinutuzumab, and venetoclax, given in combination as a treatment for CLL and/or SLL.

ELIGIBILITY:
Inclusion Criteria:

- Signed, informed consent

* Ability and willingness to comply with the requirements of the study protocol
* Age ≥18 years
* Diagnosis of the following histories according to the WHO criteria

  1. CLL or SLL
  2. MCL
* For patients with SLL, peripheral blood flow cytometry must be positive with CLL-like cells accounting for at least 1% of circulating WBC.
* No prior systemic therapy for disease under study except:

  1. prior local radiation for symptomatic disease is permitted
  2. Short course systemic corticosteroids is permissible for disease control, improvement of performance status or non-cancer indication (must be ≤ 14 days and < 100 mg/day prednisone or ≤ 20 mg/day dexamethasone). Steroids must be discontinued prior to study treatment. Inhaled steroids for asthma, topical steroids, and replacement/Stress corticosteroids are permitted. Low-dose steroids for ITP are also permitted up to the equivalent prednisone 20mg/daily at time of eligibility review.
* ECOG performance status of 0 to 2
* Adequate hematologic parameters unless due to disease under study:

  1. Absolute neutrophil count (ANC) ≥1.0 x 109/L unless neutropenia is clearly due to disease under study (per investigator discretion)
  2. Platelet count ≥ 75,000/mm3 - OR - Platelet count ≥ 20,000/mm3 if thrombocytopenia is clearly due to disease under study (per investigator discretion)
  3. Hemoglobin ≥9.0 g/dL unless anemia is clearly due to marrow involvement due to disease under study (per investigator discretion)
* Adequate renal and hepatic function, per laboratory reference range at Screening as follows:

  a. AST/SGOT, ALT/SGPT ≤2.0 x ULN b. Total bilirubin ≤ 2.0 x ULN unless:

  i. Considered secondary to Gilbert"s syndrome, in which case ≤3 x ULN ii. Considered due to disease under study (Per PI or Co-PI discretion)

  c. Creatinine clearance of eGFR>30 mL/min according to the Cockcroft-Gault Equation
* For females of childbearing potential, a negative serum pregnancy test within 7 days of study treatment
* For female patients of childbearing potential, agreement to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [<1% per year] when used consistently and correctly) or remain abstinent (refrain from heterosexual intercourse) during the treatment period and to continue its use for 90 days after the last dose of zanubrutinib AND 30 days after the last dose of venetoclax AND for 18 months after the last dose of obinutuzumab (whichever date is later)

A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (>/= 12 continuous months of amenorrhea with no identified cause other than menopause), and it not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Mullerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations.

Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Hormonal contraceptive methods must be supplemented by a barrier method.

1. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

   * For men with a female partner of childbearing potential or a pregnant female partnet: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom during the treatment period and to continue its use for 90 days after the last dose of zanubrutinib, or venetoclax AND for 18 months after the last dose of obinutuzumab (whichever date is later)

   The reliability of sexual abstinence should be evaluated in relation duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception - Willingness to not donate or bank sperm or oocytes during the entire study treatment period and after treatment discontinuation for 90 days after the last dose of zanubrutinib AND 30 days after the last dose of venetoclax AND for 18 months after the last dose of obinutuzumab (whichever date is later)

   Additional Eligibility Criteria for CLL Cohort:

   1. Diagnosis of untreated CLL or SLL according to WHO criteria 2. For patients with SLL, peripheral blood flow cytometry must be positive with CLL-like cells accounting for at least 1% of circulating WBC 3. No prior systemic therapy for CLL: prior single site of local radiation for symptomatic disease is permitted 4. Subject requires treatment according to IWCLL guidelines (See Appendix A)

   Additional Eligibility Criteria for TP53 Mutant MCL cohorts:

   1. Diagnosis of untreated stage II-IV mantle cell lymphoma

a. Prior radiotherapy for localized disease is permitted 2. Presence of TP53 mutation irrespective of variant allele frequency (TP53 cohort)

OR

Presence of p53 overexpression by immunohistochemistry defined as strong nuclear staining of >30% positive nuclei.

Additional Eligibility Criteria for Transplant Ineligible MCL cohort:

1. Diagnosis of untreated stage II-IV mantle cell lymphoma

   1. Prior radiotherapy for localized disease is permitted
2. Patients must meet one of the following criteria (a or b):

   a. Age ≥65 years If age <65 years of age, then patients must be ineligible for HDT/ASCT on the basis of comorbidity or organ dysfunction.

   Specifically, patients must meet at least one of the following criteria below:

   i.. Comorbid disease, such as CAD, CHF, pulmonary dysfunction, liver or kidney dysfunction, precluding high dose therapy secondary to expected increased morbidity and mortality. ii. ECOG 2 iii. Ejection fraction ≥35% and <45% iv. Impaired pulmonary function test with DLCO <50% expected v. Medical conditions which in the opinion of the treating physician in consultation with the study PI or Co-PI and DMT preclude HDT/ASCT.

   Exclusion Criteria:

   Other malignancies:
   * Known active histological transformation from CLL to an aggressive lymphoma (i.e., Richter"s transformation)
   * Active malignancy or systemic therapy for another malignancy within 3 years; local/regional therapy with curative intent such as surgical resection or localized radiation within 3 years of treatment is permitted
   * Other diagnosis of active cancer

   Co-morbidities:

   - Any uncontrolled illness that in the opinion of the investigator would preclude administration of study therapy (e.g. significant active infections, hypertension, angina, arrhythmias, pulmonary disease, or autoimmune dysfunction)
   * Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1, Day 1
   * Known bleeding diathesis
   * Prior major surgical procedure within 4 weeks of study, or anticipation of need for a major surgical procedure during the course of the study
   * Known CNS hemorrhage or stroke within 6 months of the study
   * History of progressive multifocal leukoencephalopathy (PML)
   * History of HIV infection

     1. Patients with a history of HIV infection that is well controlled on antiretroviral therapy are eligible if all of the following criteria are met: (1) undetectable HIV viral load by standard clinical assay AND (2) CD4+ T cell count of ≥ 200 cells/microliter

   NOTE: Many HIV regimens are excluded based on drug interactions, and concomitant antiretroviral therapy need to cleared by the clinical pharmacist and approved by the site PI)
   * Active hepatitis B (chronic or acute) or hepatitis C infection a. Patients with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV DNA is undetectable. These patients must be willing to take appropriate anti-viral prophylaxis as indicated and undergo monthly DNA testing.

     b. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
   * Congestive heart failure, New York Heart Association classification III/IV
   * Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
   * Receipt of live-virus vaccines within 28 days prior to the initiation of study treatment or need for live-virus vaccines at any time during study treatment
   * Known condition or other clinical situation that would affect oral absorption
   * Psychiatric illness/social situations that would interfere with study compliance
   * Inability to swallow a large number of tablets

   Concomitant medications and drug interactions:

   - Administration within 7 days prior to the first dose of study drug or concurrent therapy with strong inhibitors or inducers of CYP3A, CYP2C8, CYP2C9 and CYP2C19. The same applied for moderate inhibitors or inducers of CY_3A
   * Live-virus vaccines given within 28 days prior to the initiation of study treatment
   * Immunotherapy
   * Hormone therapy (other than contraceptives, hormone replacement therapy, or megestrol acetate)
   * Any therapies intended for the treatment of lymphoma/leukemia whether FDA approved or experimental (outside of this study)
   * Radiation therapy intended to treat MCL or CLL/SLL
   * Warfarin or warfarin derivatives
   * Consumption of one or more of the following within 3 days prior to the first dose of study drug:

   Grapefruit or grapefruit products Seville oranges, including marmalade containing Seville oranges Star Fruit (carambola)

   Prior therapy:
   * Prior anti-CD20 monoclonal antibody therapy for non-malignant indication
   * Obinutuzumab is contraindicated in patients with a known hypersensitivity (IgE-mediated) reaction to obinutuzumab or to any of its excipients
   * Prior systemic therapy for CLL; prior single site of local radiation for symptomatic disease is permitted

   Other:
   * Females who are currently pregnant or breastfeeding
   * Participation in a separate investigational therapeutic study unless authorized by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
establish the rate of minimum residual disease (MRD) undetectable response | 1 year
  Patients will have their minimum residual disease (MRD) response classified by bone marrow peripheral blood flow cytometry with a sensitivity of 10-4.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zelenetz, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Northwestern University, Evanston, Illinois
  - Massachusetts General Hospital (Data Collection and Specimen Analysis), Boston, Massachusetts
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- [Derived] Kumar A, Soumerai J, Abramson JS, Barnes JA, Caron P, Chhabra S, Chabowska M, Dogan A, Falchi L, Grieve C, Haydu JE, Johnson PC, Joseph A, Kelly HE, Labarre A, Lue JK, Martignetti R, Mi J, Moskowitz A, Owens C, Plummer S, Puccio M, Salles G, Seshan V, Simkins E, Slupe N, Zhang H, Zelenetz AD. Zanubrutinib, obinutuzumab, and venetoclax for first-line treatment of mantle cell lymphoma with a TP53 mutation. Blood. 2025 Jan 30;145(5):497-507. doi: 10.1182/blood.2024025563. PMID 39437708
- [Derived] Soumerai JD, Mato AR, Dogan A, Seshan VE, Joffe E, Flaherty K, Carter J, Hochberg E, Barnes JA, Hamilton AM, Abramson JS, Batlevi CL, Matasar MJ, Noy A, Owens CN, Palomba ML, Kumar A, Takvorian T, Ni A, Choma M, Friedman C, Chadha P, Simkins E, Ruiters J, Sechio S, Portman D, Ramos L, Nolet N, Mahajan N, Martignetti R, Mi J, Scorsune K, Lynch J, McGree B, Hughes S, Grieve C, Roeker LE, Thompson M, Johnson PC, Roshal M, Huang J, Biondo J, Wu Q, Jacob A, Abdel-Wahab O, Zelenetz AD. Zanubrutinib, obinutuzumab, and venetoclax with minimal residual disease-driven discontinuation in previously untreated patients with chronic lymphocytic leukaemia or small lymphocytic lymphoma: a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2021 Dec;8(12):e879-e890. doi: 10.1016/S2352-3026(21)00307-0. PMID 34826411
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm